CLINICAL TRIAL: NCT03853889
Title: Evaluation of the Effect of Epidural Anesthesia on Optic Nerve Sheath Diameter in Patients Undergoing Cesarean Section
Brief Title: Evaluation of the Effect on Optic Nerve Sheath Diameter in Patients Undergoing Cesarean Section
Acronym: EONSDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Murat Bilgi, Principal Investigator, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ABANTIBU 6
Record Dates: First submitted 2019-01-11; First posted 2019-02-26 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Intracranial Pressure
Keywords: optic nerve sheath pressure; noninvasive intracranial pressure measurement; epidural anesthesia; cesarean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preepidural ONSD (Active Comparator): The diameter of the optic nerve sheath to be measured(ONSD) with the help of ultrasonography before epidural anesthesia(pre epidural ONSD). The measurement will be measured 3 mm behind the optical disc. The measurements shall be applied in both transverse and sagittal planes for both eyes and the arithmetic mean of the four measured values.
  Interventions: Procedure: USG guided ONSD measurement preepidural
- post epidural ONSD (Experimental): The diameter of the optic nerve sheath to be measured with the help of ultrasonography Immediately after epidural anesthesia(post epidural ONSD) (T1), 15 minutes (T2), 30 min (T3), 60. min (T4) epidural anesthesia. The measurement will be measured 3 mm behind the optical disc. The measurements shall be applied in both transverse and sagittal planes for both eyes and the arithmetic mean of the four measured values.
  Interventions: Procedure: USG guided ONSD measurement preepidural

INTERVENTIONS:
Procedure: USG guided ONSD measurement preepidural — Measurement of the diameter of the optic nerve sheath preepidural and postepidural anesthesia
  Other Names: USG guided ONSD measurement postepidural

SUMMARY:
Depending on the physiology of pregnancy, the risk of increased aspiration, difficult airway, increased oxygen consumption and reduced functional residual capacity, breathing problems make general anesthesia application risky. In obstetric operations, neuraxial anesthesia is preferred because of both maternal and maternal mortality and morbidity. Epidural area has decreased due to pregnancy physiology. Previous studies have shown that the blood given to the epidural area increases the intracranial pressure by compressing the dura mater.Optic nerve diameter measurements ultrasound guided is a non-invasive and reliable method for detecting intracranial pressure increase.

In this study, aimed to compare the optic nerve sheath diameter before and after epidural anesthesia with USG.

DETAILED DESCRIPTION:
Epidural anesthesia will be performed at L2 level and sitting position in all patients. Patients will be measured and recorded for optic nerve sheath diameter at 15 min (T2), 30 min (T3) and 60 min (T4) immediately after epidural anesthesia (T0) and after epidural anesthesia.. Measurement of the optic nerve sheath diameter will be done with the help of a linear probe without applying high pressure to the eyeball while the patient is in supine position and the eyelids are closed. The optic nerve sheath diameter will be measured 3 mm beyond the optical disc. The measurements shall be applied in both transverse and sagittal planes for both eyes and the arithmetic mean of the four measured values.

ELIGIBILITY:
Inclusion Criteria:

* epidural anesthesia patients
* 18-40 years patients
* American Society of Anesthesiologists status I-II patients

Exclusion Criteria:

* Patients with allergy to any of the drugs to be used in the study,
* patients with severe heart failure,
* atrial and ventricular arrhythmias,
* severe valve disease,
* electrolyte disorder,
* renal failure, preeclampsia, eclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-06-28 (Estimated); Primary Completion 2019-08-17 (Estimated); Study Completion 2019-12-17 (Estimated)

PRIMARY OUTCOMES:
increase in the diameter of the optic nerve sheath after epidural anesthesia | Basal(T0),Immediately after administration of epidural anesthesia(T1), after epidural anesthesia 15 min(T2), 30 min (T3),60 min (T4)
  increase of intracranial pressure as a result of the administration of 20 ml of local anesthetic to the epidural area and its reflection on the diameter of the optic nerve sheath

CONTACTS AND LOCATIONS:
Overall Officials: murat bilgi, MD, Principal Investigator — Bolu Abant İzzet Baysal University